CLINICAL TRIAL: NCT01379378
Title: Male Stress Urinary Incontinence and Sexual Health
Status: Withdrawn | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: PROS0035; SU-06152011-7928 (Other: Stanford University)
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Urinary Sphincter, Artificial; glutaraldehyde-cross-linked collagen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Artificial urinary sphincter — Standard of care
  Other Names: urethral sphincter; American Medical Systems
Device: InVance Sling — Standard of care
  Other Names: Urithrary sling; American Medical Systems
Device: AdVance Sling — Standard of care
  Other Names: Urithrary sling
Device: Virtue Sling — Standard of care
  Other Names: Coloplast
Drug: Contigen — 2.5-10 cc
  Other Names: Bard

SUMMARY:
The purpose of this study if to demonstrate if post-prostatectomy incontinence is a barrier to sexual satisfaction/frequency/desire and if surgical correction of incontinence will improve these aspects of sexual health.

ELIGIBILITY:
Inclusion Criteria:

* Adult men age 18-80 who have had an open or laparoscopic radical prostatectomy more than 6 months ago who have bothersome urinary incontinence.

Exclusion Criteria:

* Any significant cardiac or pulmonary co-morbidities that would preclude the patient from another surgical procedure as they would be too high risk for general anesthesia.
* They will also be excluded if based on their anatomy or urodynamics, they will most likely not benefit from a surgical incontinence procedure (e.g. poor bladder contractility, bladder neck contracture, etc).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-prostatectomy patients at least 6 months after either open radical retropubic prostatectomy or robot assisted laparoscopic prostatectomy with bothersome stress urinary incontinence will be initially screened with urodynamics, a 24 hour pad test, and a self questionnaire to assess how bothersome their incontinence is.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Whether stress urinary incontinence is a barrier to sexual satisfaction/frequency/desire | 1 year
Whether surgical correction of stress urinary incontinence will improve these aspects of sexual health | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Craig Vance Comiter, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States